CLINICAL TRIAL: NCT00743574
Title: Health Benefits of Vitamin D and Calcium in Women With PCOS (Polycystic Ovarian Syndrome)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YaleU-0807003992; YCCI-CARE Grant #UL1RR024139
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Results first posted 2013-07-29 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovarian Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency | interventions — Ergocalciferols; Medroxyprogesterone; Medroxyprogesterone Acetate; Cholecalciferol; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D plus Calcium (Ca) supplementation (Experimental)
  Interventions: Dietary Supplement: Vitamin D2 (Ergocalciferol); Drug: Medroxyprogesterone (Provera); Dietary Supplement: Vitamin D3 (Cholecalciferol); Dietary Supplement: Elemental Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D2 (Ergocalciferol) — 50,000IU (or 1 tablet), PO, monthly (supplements to be taken for three months)
Drug: Medroxyprogesterone (Provera) — 10mg, PO, daily for ten days
Dietary Supplement: Vitamin D3 (Cholecalciferol) — 2,000IU (or 2 tablets), PO, daily (supplements taken for three months)
Dietary Supplement: Elemental Calcium — 1,000mg (or 2 tablets), PO, daily (supplements taken for three months)

SUMMARY:
The investigators conducted a prospective un-blinded pilot study of Vitamin D plus Calcium (Ca) supplementation in overweight (BMI > 27) premenopausal women diagnosed with Polycystic Ovarian Syndrome (PCOS), as defined by the Rotterdam Criteria, 2003, and who were deficient in vitamin D as reflected by serum 25-hydroxy (25-OH) vitamin D (serum levels < 20 ng/mL).

DETAILED DESCRIPTION:
We had hypothesized that in women with PCOS, administering optimal daily doses of vitamin D3, as recommended by the National Academy of Sciences, 2000IU Cholecalciferol and 1000mg of calcium, both per oral (PO), over a three month period will improve their metabolic picture, and possibly hormone profile.

Over the course of the trial, after the first 5 subjects had completed 3 month intervention,we observed that daily 2000IU D3 dosing regime was inadequate in normalizing vitamin D status in the study population; the dosing regimen was therefore modified to include weekly supplementation with 50,000IU D2 in addition to daily dosing with 2000IU D3.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women (ages 18-40 years) with normal thyroid function and prolactin levels.
* PCOS diagnosis based on Rotterdam criteria: presence of at least 2 of the following criteria:

  * oligomenorrhea-menstrual cycles > 35 day intervals
  * hyperandrogenemia (elevated serum testosterone [free or total] &/or androstenedione levels) or features of hyperandrogenism i.e. acne or hirsuitism [Ferriman-Gallaway score > 3]
  * polycystic ovaries on vaginal ultrasound as defined by ESHRE/ASRM criteria (ovarian volume ≥ 10mL or ≥ 12 follicles of diameter between 2-9mm in at least one ovary)
  * Overweight (BMI ≥ 27 Kg/m2)
  * Biochemical evidence of Vitamin D insufficiency (i.e. serum 25 OHD levels < 20ng/mL)

Exclusion Criteria:

* Pregnancy
* Known causes of oligomenorrhea other than PCOS, e.g. hypothyroidism/Cushing's Disease/late onset congenital adrenal hyperplasia (fasting 17-alphahydroxyprogesterone levels < 200ng/dL)
* Use of hormonal treatment (birth control pill/patch/depot medroxyprogesterone/medroxyprogesterone) within 3 months of the study onset.
* Use insulin sensitizers (metformin, sulfonylureas, TZDs, incretins) within 3 months of the study onset.
* Use of lipid lowering agents or medications known to influence insulin sensitivity (e.g. niacin, corticosteroids, beta blockers, calcium channel blockers, thiazide diuretics) or influence serum androgens (estrogen, anti-androgens, androgens) within 3 months of the study onset.
* Known history of renal calculi or current use of Calcium and Vitamin D supplements.
* Spanish Speaking.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lubna Pal, MBBS,MRCOG,MSc., Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital-Women's Center, New Haven, Connecticut, United States

REFERENCES:
- [Result] Pal L, Berry A, Coraluzzi L, Kustan E, Danton C, Shaw J, Taylor H. Therapeutic implications of vitamin D and calcium in overweight women with polycystic ovary syndrome. Gynecol Endocrinol. 2012 Dec;28(12):965-8. doi: 10.3109/09513590.2012.696753. Epub 2012 Jul 11. PMID 22780885
- [Derived] Nardell M, Chhabra A, Pal L. Excluded, not dismissed: enhancing benefit in clinical research. Contemp Clin Trials. 2013 Jan;34(1):70-3. doi: 10.1016/j.cct.2012.08.013. Epub 2012 Sep 7. PMID 22981957

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited through flyers, medical clinics, internet postings May 2008-February 2010
Pre-assignment Details: Some subjects did not follow through with eligibility testing or had further exclusions, such as scheduling difficulties.
Groups:
- Vitamin D Plus Calcium (Ca) Supplementation: Vitamin D3 (Cholecalciferol) : 2,000IU (or 2 tablets), PO, daily (supplements taken for three months)
  Elemental Calcium : 1,000mg (or 2 tablets), PO, daily (supplements taken for three months)
  Vitamin D2 (Ergocalciferol) : 50,000IU (or 1 tablet), PO, monthly (supplements to be taken for three months)
  Medroxyprogesterone (Provera) : 10mg, PO, daily for ten days
Period: Overall Study
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Started | 36
Dropped Out Before Eligibility Testing | 13
Further Exclusions | 8
Dropped Out After Initiating Trial | 3
Completed | 12
Not Completed | 24

BASELINE CHARACTERISTICS:
Population: the number of participants for analysis was determined by the number who completed the study.
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.42 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Baseline HbA1C levels [Mean (Standard Deviation); unit: percentage] — Fasting HbA1C levels were collected at baseline during a 2 hour oral Glucose Tolerance Test (GTT)
  percentage | 5.37 (0.53)
Baseline insulin levels [Mean (Standard Deviation); unit: µIU/ml] — Fasting insulin levels at baseline were drawn during an oral GTT
  µIU/ml | 24.92 (15.42)
Baseline glucose levels [Mean (Standard Deviation); unit: mg/dl] — Fasting glucose levels at baseline were drawn during an oral GTT
  mg/dl | 103.79 (22.83)
Baseline AUC insulin [Mean (Standard Deviation); unit: µIU/ml/120 min] — Fasting AUC (Area under the curve at 0, 0.5, 1, 1.5 and 2 hours)insulin was drawn at baseline during a oral GTT
  µIU/ml/120 min | 16136.50 (10086.29)
Baseline AUC for glucose [Mean (Standard Deviation); unit: mg/min/120min] — Fasting level for AUC (Area under the curve at 0, 0.5, 1, 1.5 and 2 hours)glucose at baseline was drawn based on oral GTT
  mg/min/120min | 16648.41 (3949.98)
Baseline C Reactive protein level [Median (Inter-Quartile Range); unit: mg/L] — Fasting levels of Creactive protein levels were drawn during oral GTT
  mg/L | 5.72 (1.51-13.93) [1.51 to 13.93]

OUTCOME MEASURES:

1. Secondary Outcome: Serum Levels of C-reactive Protein at Completion of 3 Months Treatment
Description: Serum levels of C-reactive protein upon completion, at 3 months
Time Frame: 3 months
Population: All subjects who completed treatment for 3 months
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
mg/L | 5.3 [1.52 to 14.36]

2. Primary Outcome: Serum HbA1C at 3 Months
Description: Fasting HbA1C levels at study completion after 3 month treatment
Time Frame: Completion
Population: Number determined by those who completed all interventions and procedures.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
percentage | 5.55 (0.66)

3. Primary Outcome: Fasting Insulin Levels at Study Completion After 3 Month Treatment
Description: Fasting insulin levels at study completion after 3 month treatment
Time Frame: 3 months intervention
Population: Number determined by all those who completed all interventions and procedures.
Measure: Mean (Standard Deviation); unit: µIU/ml
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
µIU/ml | 25.17 (13.67)

4. Primary Outcome: Fasting Glucose Levels at Completion of Treatment, at 3 Months
Description: Fasting glucose levels drawn after 3 months completion during oral GTT
Time Frame: 3 months
Population: Number determined based on all interventions and procedures completed.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
mg/dl | 103.79 (22.83)

5. Primary Outcome: AUC (Area Under a Curve at 0, 0.5, 1, 1.5 and 2 Hours) Insulin During 2 Hour GTT at Completion, at 3 Months
Description: Following 3 months intervention, AUC insulin was determined during 2 hour oral GTT
Time Frame: 3 months
Population: Number determined by completion of all study interventions and procedures
Measure: Mean (Standard Deviation); unit: µIU/ml/120min
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
µIU/ml/120min | 16715.57 (10371.76)

6. Primary Outcome: AUC (Area Under the Curve at 0, 0.5, 1, 1.5 and 2 Hours) During Oral GTT at Completion, at 3 Months
Description: AUC (Area under the curve at 0, 0.5, 1, 1.5 and 2 hours)for glucose was determined at completion of 3 months intervention for 2 hour oral GTT
Time Frame: 3 months
Population: Number determined by all participants who completed all interventions and procedures
Measure: Mean (Standard Deviation); unit: mg/min/120min
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Number analyzed (Participants) | 12
mg/min/120min | 16726.56 (3941.80)

ADVERSE EVENTS:
Arm/Group | Vitamin D Plus Calcium (Ca) Supplementation
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
No limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes